CLINICAL TRIAL: NCT05226234
Title: Risk Stratification of VT / VF After Myocardial Infarction Based on Cardiac MRI 2
Acronym: TVScreen-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Christian DE CHILLOU, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2021PI063
Record Dates: First submitted 2022-01-17; First posted 2022-02-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Myocardial Infarction; Ventricular Tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Myocardial Infarction; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Late gadolinium enhancement cardiac magnetic resonance (LGE-MRI)

SUMMARY:
Implantable cardioverter-defibrillators (ICD) are currently recommended (ESC guidelines 2015) for the primary prevention of sudden cardiac death (SCD) in patients with a remote myocardial infarction (MI) and a low (≤35%) left ventricular ejection fraction (LVEF). Ventricular tachycardia (VT) and/or ventricular fibrillation (VF), which are responsible for most SCDs, result from the presence of surviving myocytes embedded within fibrotic MI-scar. The presence of these surviving myocytes, as well as their specific arrhythmic characteristics, is not captured by LVEF. Consequently, most patients with a prophylactic ICD do not present VT/VF requiring ICD therapy prior to their first-ICD battery depletion. Thus, many patients are exposed to ICD complications, such as inappropriate shocks, without deriving any health benefit. As a consequence, the current implantation strategy of prophylactic ICDs, based on LVEF, needs to be improved in post-MI patients. Stratification of the rhythmic risk after IDM is therefore still a major public health issue.

Late gadolinium enhancement cardiac magnetic resonance (LGE-MRI) is a strong risk-stratifier of VT/VF risk in post- MI patients. In a recent multicenter retrospective study, the investigators showed that the presence of a critical surface of intramural scar (which is consequently neither epicardial nor endocardial) at the infarct border (measured by LGE-MRI) has a major association with the occurrence of VT/VF in post-MI patients with a LVEF≤35%.

The aim of the TVScreen 2 study is therefore to validate the relevance of the MRI criterion in a new independent cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Person who has received full information on the organization of the research and who has not objected to the use of this data;
* Person having had an ICD implantation for primary prevention before 12/31/2017 after myocardial infarction;
* Person with LVEF ≤35% at the time of ICD implantation.

Exclusion Criteria:

* Patient with a history of persistent atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of myocardial infarction with LVEF ≤35%, implantation of an ICD for primary prevention before 12/31/2017 and the performance of a cardiac MRI.
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between the presence of the MRI criterion "intramural scar ≥ 1.47cm²" measured by MRI and the occurrence of VT / VF after implantation of the ICD from the patient's medical record. | 5 years
  The area of the intramural scar will be determined from the MRI images. VT / VF events during the follow-up period will be reported from cardiac events recorded by the ICD and present in the patient's medical record.

SECONDARY OUTCOMES:
Association between the MRI criterion "intramural scar ≥ 1.47cm²" measured by MRI and all-cause mortality from the patient's medical record. | 5 years
  The area of the intramural scar will be determined from the MRI images. All-cause mortality during the follow-up period will be collected from the patient's medical record.
Association between the MRI criterion "intramural scar ≥ 1.47cm²" measured by MRI and the combined criterion of all-cause mortality or occurrence of VT / VF from the patient's medical record. | 5 years
  The area of the intramural scar will be determined from the MRI images. VT / VF events and all-cause mortality during the follow-up period will be collected as described previously.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France